CLINICAL TRIAL: NCT01540474
Title: Phase 1 Study With the Vaccine Candidate Plasmodium Falciparum Malaria Protein (FMP012), an E.Coli-expressed Cell-Traversal Protein, Administered Intramuscularly in Healthy Malaria-Naive Adults
Brief Title: Trial of a Falciparum Malaria Protein (FMP012), E. Coli-expressed PfCelTOS, in Healthy Malaria-Naive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-11-21; IND 014962 (Other: WRAIR)
Record Dates: First submitted 2012-02-09; First posted 2012-02-28 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Malaria
Keywords: Interference of malaria infection
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: 10 ug FMP012 with 2 ug GLA-SE (Experimental): Single center, non-randomized, open label, dose escalation Phase 1 study with sporozoite challenge. The antigen FMP012 will be adjuvanted with Glucopyranosyl lipd A stable emulsion. This is a first-in-human study of FMP012. 30 subjects, divided into 3 groups, will receive 3 doses of the FMP012/GLA-SE vaccine. Biological/vaccine; E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipid A Stable emulsion (GLA-SE), a proprietary adjuvant
  Interventions: Biological: Group 1: 10 ug FMP012 with 2 ug GLA-SE
- Group 2: 10 ug FMP012 with 5 ug GLA-SE (Experimental): Biological/vaccine; E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipid A Stable emulsion (GLA-SE), a proprietary adjuvant
  Interventions: Biological: Group 2: 10 ug FMP012 with 5 ug GLA-SE
- Group 3: 50 ug FMP012 with 5 ug GLA-SE or 2 ug GLA-SE (Experimental): Biological/vaccine; E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipid A Stable emulsion (GLA-SE), a proprietary adjuvant
  Interventions: Biological: 50 ug FMP012 with 5 ug GLA-SE or 2 ug GLA-SE
- Control group-Challenged Only (Other): Biological/vaccine; E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipid A Stable emulsion (GLA-SE), a proprietary adjuvant
  Interventions: Other: Controlled group-Challenged Only: no vaccination

INTERVENTIONS:
Biological: Group 1: 10 ug FMP012 with 2 ug GLA-SE — Biological/vaccine; E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipid A Stable emulsion (GLA-SE), a proprietary adjuvant
  Arms: Group 1: 10 ug FMP012 with 2 ug GLA-SE
Biological: Group 2: 10 ug FMP012 with 5 ug GLA-SE — E-coli expressed antigen FMP012 will be adjuvanted with Glucopyranosyl lipd A stable emulsion (GLA-SE), a proprietary adjuvant
  Arms: Group 2: 10 ug FMP012 with 5 ug GLA-SE
Biological: 50 ug FMP012 with 5 ug GLA-SE or 2 ug GLA-SE — E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipd A stable emulsion (GLA-SE), a proprietary adjuvant
  Arms: Group 3: 50 ug FMP012 with 5 ug GLA-SE or 2 ug GLA-SE
Other: Controlled group-Challenged Only: no vaccination — The control group participated in the primary malaria sporozoite challenge.E-coli expressed antigen FMP012 will be adjuvanted with Glucopyranosyl lipd A stable emulsion (GLA-SE), a proprietary adjuvant
  Arms: Control group-Challenged Only

SUMMARY:
Malaria has remained a major concern for the US military. During World War II, malaria was the leading cause of disease and non-battle injury with 500-700 men infected per day, resulting in 24,000 malaria-related casualties.(10) Currently, the methods used for protecting troops against malaria are insecticidal nets, clothing, and antimalarial treatment. To be effective, these methods must be self-administered and be used consistently, often unattainable in field or combat situations. The United States Army Medical Research and Development Command (USAMRMC), through the United States Army Medical Materiel Development Activity (USAMMDA) and the Walter Reed Army Institute of Research (WRAIR) are actively pursuing the development of an effective vaccine against P. falciparum malaria; development of such a vaccine is a high priority for the US military and other individuals who travel to endemic regions, and is equally important to populations residing in those areas.

A Phase 1 study using FMP012, a recombinant E.coli expressed malaria protein (CelTOS) vaccine will

1. assess the safety and reactogenicity of candidate P. falciparum malaria vaccine FMP012/GLA-SE

   Secondary:
2. measure the humoral immune response to FMP012/GLA-SE using enzyme-linked immunosorbent assay (ELISA)
3. assess the protective efficacy of FMP012/GLA-SE against a P. falciparum sporozoite challenge.

DETAILED DESCRIPTION:
Single center, non-randomized, open label, dose escalation Phase 1study with sporozoite challenge. The antigen FMP012 will be adjuvanted with Glucopyranosyl lipd A stable emulsion (GLA-SE), a proprietary adjuvant produced by the Infectious Disease Research Institute (IDRI). This is a first-in-human study of FMP012. Thirty subjects, divided into 3 groups (10 subjects per group), will receive 3 doses of the FMP012/GLA-SE vaccine. Group 1 will receive 10 µg of FMP012 formulated with 2 µg GLA-SE adjuvant and Group 2 will receive 10 µg of FMP012 formulated with 5 µg GLA-SE adjuvant. Group 3 will receive 50 µg of FMP012 formulated with either 5 µg GLA-SE adjuvant (Group 3a) or 2 µg GLA-SE adjuvant (Group 3b). Determination of whether to proceed with Group 3a or Group 3b will be made by the principal investigator (PI) and the independent medical monitor after the second vaccination dose in Group 2 has been completed, based on predefined safety and group hold criteria in this protocol. There will be a staggered start for Group 1 and Group 2 separated by a minimum of 14 days. Group 3a or Group 3b will start vaccinations 2 weeks after the second vaccination for Group 2. The first and second vaccination doses in each group will be separated by 28 days and all groups will receive the third vaccination dose on the same day. The second and third vaccination doses in Group 1 will be separated by 84 days, Group 2 by 70 days, and Group 3 by 28 days. Six non-immunized infectivity control subjects will be enrolled prior to the challenge phase. All subjects from the Vaccination Group and Infectivity Control Group will participate in the primary malaria sporozoite challenge and will be required to stay at a hotel for evaluation for a maximum of 10 nights starting 9 days after the challenge. A directly monitored, sequentially allocated, open-label oral regimen of chloroquine or artemether/lumefantrine will be administered to all parasitemic subjects.

ELIGIBILITY:
* Healthy adults (male or non-pregnant, non-lactating female) 18 to 50 years of age at the time of screening
* If the subject is female,
* Non-childbearing potential , abstinent or using adequate contraceptive precautions during this study and must agree to continue such precautions until three months after challenge
* A negative pregnancy test at the time of enrollment
* Free of significant health problems as established by medical history, laboratory, and clinical examination before entering the study
* Low cardiac risk factors
* Available to participate and reachable by phone for duration of study (approximately 8 months)
* No plans to travel to outside the Washington DC area between the day of challenge and either completion of treatment course (post-challenge) or, if subject remains uninfected, 28 days post-challenge
* No plans to travel to a malaria endemic area during the course of the study
* Written informed consent must be obtained from the subject before screening procedures
* Subjects must score at least 80% correct on a multiple-choice quiz that assesses their understanding of this study
* Active duty military must obtain approval from his or her supervisor

Exclusion Criteria:

* History of malaria infection
* History of travel to P. falciparum endemic areas in the 3 months prior to day of first vaccination or day of challenge
* History of receiving a malaria vaccine
* Receipt of any licensed vaccine within 7 days prior to first vaccination
* History of receipt of malaria prophylaxis during the 2 months prior to day of first vaccination or day of challenge
* History of use of any drugs with significant antimalarial activity during the course of the study period
* Prior receipt of any vaccine containing either QS-21, MPL or GLA-SE in the previous 5 years (including Cervarix®, GSK)
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine or planned use during the study period.
* Any history of allergic reaction or anaphylaxis to previous vaccination
* Allergy to kanamycin, nickel, or imidazole Pregnant or lactating female at screening or plans to become pregnant or breastfeed from the time of enrollment until three months after challenge
* Allergy to antimalarial drugs or use of medications known to interact with both CQ and artemether/lumefantrine
* Significant (eg, systemic) hypersensitivity reactions to mosquito bites
* History of sickle cell disease
* History of psoriasis or porphyria
* History of splenectomy
* Any confirmed or suspected immunodeficiency, including HIV infection
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune-modifying drugs within six months of vaccination
* Inhaled and topical steroids are allowed
* A family history of congenital or hereditary immunodeficiency
* Acute or chronic, clinically significant, pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by history, physical examination, or laboratory evaluation
* Chronic or active neurologic disease including seizure disorder and chronic migraine headaches
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or any planned administration during the study period
* Any abnormal baseline laboratory screening tests listed below (normal values are defined in the adverse event section of this protocol):
* Seropositive for HIV or Hepatitis C virus or HBsAg positive
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* An abnormal baseline screening EKG.
* Suspected or known current alcohol or drug abuse as determined from the medical history or by physical examination
* Any other significant finding that in the opinion of the PI would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica J. Cowden, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Clinical Trials Center, WRAIR, Silver Spring, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Infectivity Controls participating in the study at the challenge stage; no vaccinations received or placebos prior to the challenge
Period: Vaccination Period
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
Started | 10 | 10 | 10 | 0
Completed | 10 | 9 | 10 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Malaria Challenge
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
Started | 10 | 9 | 10 | 6
Completed | 10 | 9 | 10 | 5
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group | Total
Number analyzed (Participants) | 10 | 10 | 10 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (8.37) | 31.1 (10.17) | 34.3 (10.88) | 28.3 (8.41) | 32.4 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 3 | 2 | 13
  Male | 7 | 5 | 7 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 9 | 10 | 6 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 2 | 1 | 10
  White | 7 | 5 | 6 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Active Duty [Count of Participants; unit: Participants] | 4 | 1 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited or Unsolicited Symptoms Reporting During the Post-vaccination Period
Description: Number of participants for each dose (1 through 3) that experienced any symptom, general solicited symptoms, and local solicited symptoms
Time Frame: From vaccination day through 7 days post vaccination (for all three doses)
Population: Three dosing groups vaccinated with three doses of vaccine at varying intervals + an infectivity control group (malaria challenge phase only)
Measure: Number; unit: participants
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
Number analyzed (Participants) | 10 | 10 | 10 | 0
participants
  Any Symptoms Dose 1 | 10 | 10 | 9 |
  Any Symptom Dose 2 | 10 | 10 | 9 |
  Any Symptom Dose 3: number analyzed (Participants) | 10 | 9 | 10 | 0
  Any Symptom Dose 3 | 8 | 9 | 4 |
  General Solicited Symptoms Dose 1 | 3 | 5 | 1 |
  General Solicited Symptoms Dose 2 | 3 | 3 | 3 |
  General Solicited Symptoms Dose 3: number analyzed (Participants) | 10 | 9 | 10 | 0
  General Solicited Symptoms Dose 3 | 0 | 1 | 0 |
  Local Solicited Symptoms Dose 1 | 9 | 10 | 9 |
  Local Solicited Symptoms Dose 2 | 8 | 9 | 9 |
  Local Solicitied Symptoms Dose 3: number analyzed (Participants) | 10 | 9 | 10 | 0
  Local Solicitied Symptoms Dose 3 | 10 | 9 | 10 |
  Overall/Dose Any Symptom | 28 | 29 | 22 |
  Overall/Dose General Solicited Symptoms | 6 | 9 | 4 |
  Overall/Dose Local Solicited Symptoms | 25 | 28 | 22 |
  Overall/Subject Any Symptom | 10 | 10 | 9 |
  Overall/Subject General Solicited Symptoms | 5 | 5 | 3 |
  Overall/Subject Local Solicited Symptoms | 9 | 10 | 9 |

2. Primary Outcome: Number of Participants With Solicited or Unsolicited Symptoms Reporting During the Post-vaccination Period
Description: Incidence of erythema and pain (solicited local symptoms) reported after each dose (1-3) of vaccination. Results for groups 1, 2 and 3 only as control group did not receive any vaccinations and only participated in the malaria challenge portion of the study.
Time Frame: From vaccination day through 7 days post vaccination for each does (1-3)
Population: Vaccination group only; control group participated in malaria challenge only
Measure: Number; unit: participants
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
Number analyzed (Participants) | 10 | 10 | 10 | 0
participants
  Dose 1 : Erythema All | 0 | 0 | 0 |
  Dose 1 : Erythema > 100mm | 0 | 0 | 0 |
  Dose 1 : Pain All | 9 | 10 | 9 |
  Dose 1 : Pain Grade 3 | 0 | 0 | 0 |
  Dose 2 : Erythema All | 1 | 1 | 0 |
  Dose 2 : Erythema > 100mm | 0 | 0 | 0 |
  Dose 2 : Pain All | 7 | 9 | 9 |
  Dose 2 : Pain Grade 3 | 0 | 0 | 0 |
  Dose 3 : Erythema All: number analyzed (Participants) | 10 | 9 | 10 | 0
  Dose 3 : Erythema All | 1 | 0 | 0 |
  Dose 3 : Erythema > 100mm | 0 | 0 | 0 |
  Dose 3 : Pain All | 8 | 9 | 4 |
  Dose 3 : Pain Grade 3 | 0 | 0 | 0 |
  Overall/Dose Erythema All | 2 | 1 | 0 |
  Overall/dose Erythema >100mm | 0 | 0 | 0 |
  Overall/Dose Pain All | 24 | 28 | 22 |
  Overall/Dose Pain Grade 3 | 0 | 0 | 0 |
  Overall/Subject Erythema All | 2 | 1 | 0 |
  Overall/Subject Erythema >100mm | 0 | 0 | 0 |
  Overall/Subject Pain All | 9 | 10 | 9 |
  Overall/Subject Pain Grade 3 | 0 | 0 | 0 |

3. Primary Outcome: Subjects Reporting the Occurrence of Unsolicited Adverse Events Related to Vaccination
Description: Number of participants with at lease one administered dose presenting with at least one specified symptom within 28 days after vaccination
Time Frame: 28 days after each vaccination
Population: Three dosing groups. Control group only participated in the malaria challenge portion of the study and was not vaccinated.
Measure: Number; unit: participants
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
Number analyzed (Participants) | 10 | 10 | 10 | 0
participants
  At Least 1 Symptom | 2 | 2 | 1 |
  General Disorders and Admin. Site Conditio | 2 | 1 | 1 |
  Injection Site Haemorrhage | 1 | 0 | 1 |
  Injection Site Haematoma | 0 | 1 | 0 |
  Injection Site Pruritus | 1 | 0 | 0 |
  Nervous System Disorders | 0 | 1 | 0 |
  Dizziness | 0 | 1 | 0 |

4. Secondary Outcome: Humoral Immune Response to FMP012/GLA-SE
Description: Seroconversion was defined as a post-second vaccination titer (serum dilution of 1:100) that is 3 standard deviations higher than the average of the negative or pre-vaccination serum measured using enzyme-linked immunosorbent assay (ELISA). Values reported as "below the detection limit" were given a value of 50 units. The safety population was used for immunogenicity analysis. Only subjects who received vaccinations or were challenged were included in the analysis of immunogenicity. Subjects who withdrew from the study had data collected to the point of withdraw.
  Geometric mean titers (GMT) were obtained by first calculating the mean and 95% confidence intervals for log-transformed values of the ELISA results, followed by exponentiation of the values. Among those vaccinated, all values were below the detection limit until post-dose II.
Time Frame: Up to 1 year
Population: Only subjects who received vaccinations or were challenged were included in the analysis of immunogenicity. Subjects who withdrew from the study had data collected to the point of withdraw.
Measure: Geometric Mean (95% Confidence Interval); unit: antibody titer
Groups:
- Group 3a: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE: Biological/vaccine; E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipid A Stable emulsion (GLA-SE), a proprietary adjuvant
  50 ug FMP012 with 5 ug GLA-SE: E-coli expressed malaria antigen FMP012 adjuvanted with Glucopyranosyl lipd A stable emulsion (GLA-SE), a proprietary adjuvant
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3a: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
Number analyzed (Participants) | 10 | 10 | 10 | 6
antibody titer
  Post Dose II: number analyzed (Participants) | 10 | 10 | 10 | 0
  Post Dose II | 1780.1 [685.8 to 4620.7] | 2755.5 [1041.1 to 7292.7] | 3846.6 [1352.0 to 10943.7] |
  Pre Dose III: number analyzed (Participants) | 10 | 9 | 10 | 0
  Pre Dose III | 362.9 [145.8 to 903.4] | 518.9 [180.9 to 1488.9] | 2151.9 [609.4 to 7598.9] |
  Post Dose III: number analyzed (Participants) | 10 | 9 | 10 | 0
  Post Dose III | 9503.1 [4420.9 to 20427.4] | 11110.2 [5681.6 to 21725.4] | 6744.3 [2337.7 to 19457.2] |
  Post Challenge: number analyzed (Participants) | 10 | 9 | 10 | 6
  Post Challenge | 6440.0 [2715.8 to 15271.4] | 4289.4 [2027.7 to 9074.1] | 3566.8 [1214.1 to 10478.4] | 65.2 [33.0 to 128.7]
  Final Visit: number analyzed (Participants) | 10 | 9 | 10 | 6
  Final Visit | 3077.4 [1202.6 to 7874.9] | 2099.8 [823.4 to 5354.8] | 1483.6 [499.0 to 4410.8] | 67.4 [31.3 to 145.2]

5. Secondary Outcome: Time to Onset of Parasitemia Following Sporozoite Challenge
Description: Protective Efficacy of FMP012/GLA-SE Measured against a P falciparum sporozoite challenge. Vaccinated subjects were compared to infectivity controls to assess for delayed onset of parasitemia. Time of onset of parasitemia was based on the date of sporozoite challenge to the date of first positive blood smear detection.
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3a: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
Number analyzed (Participants) | 10 | 9 | 10 | 6
days | 13.0 (0.82) | 14.6 (2.30) | 13.5 (0.85) | 14.0 (1.00)

ADVERSE EVENTS:
Time Frame: Unsolicited AEs collected through day 28 after each vaccination; SAEs collected from Day 0 through Day 225
Arm/Group | Group 1: 10 ug FMP012 With 2 ug GLA-SE | Group 2: 10 ug FMP012 With 5 ug GLA-SE | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 10 ug FMP012 With 2 ug GLA-SE (N=10) | Group 2: 10 ug FMP012 With 5 ug GLA-SE (N=10) | Group 3: 50 ug FMP012 With 5 ug GLA-SE or 2 ug GLA-SE (N=10) | Control Group (N=6)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Abdominal Cramping
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 3 (3) | 3 (3) | 1 (1) — Increased ALT
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — Right Shoulder Ache
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Insect Bite Left Thigh
Aspartate Aminotransferase Increased (Investigations) | 4 (4) | 4 (4) | 3 (3) | 2 (2) — Increased AST
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) — Low Back Pain
Blood Creatinine Increased (Investigations) | 1 (2) | 2 (2) | 0 (0) | 1 (1) — Increased Creatinine
Blood Pressure Systolic Increased (Investigations) | 0 (0) | 2 (5) | 1 (2) | 2 (4) — Elevated Systolic Blood Pressure
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Episodic Sternal Pain X 3
Chills (General disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (4) — Anorexia
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Intermittent Loose Stools
Dizziness (Nervous system disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) — Lightheadedness/Dizziness
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Allergic reaction to Artemether/Lumefantrine
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Menstrual Cramps
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Indigestion
Fatigue (General disorders) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Feeling Hot (General disorders) | 1 (2) | 2 (5) | 0 (0) | 2 (3) — Feverish (Subjective)
Food Poisening (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 3 (4) | 1 (3) | 3 (4) | 2 (3)
Headache (Nervous system disorders) | 6 (8) | 6 (25) | 4 (5) | 2 (6)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hot Flash
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Inflammatory Reaction at the Right Challenge Site
Injection Site Haemorrhage (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Ecchymosis at Right Arm Injection Site
Injection site Pain (General disorders) | 9 (24) | 10 (28) | 9 (22) | 0 (0)
Malaise (General disorders) | 3 (4) | 4 (7) | 1 (3) | 0 (0) — Fatigue/Malaise
Malaria (Infections and infestations) | 10 (10) | 9 (9) | 10 (10) | 5 (5) — Malaria Symptoms
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (3) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Sore Throat
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Sore Feet
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — 5 small papules right forearm
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) — Tingling
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Petechia around eyes
Platelet Count Decreased (Investigations) | 8 (9) | 3 (3) | 4 (4) | 2 (2)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pelvic Pain
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Vasovagal Reaction During Blood Draw
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 4 (4) | 2 (3) | 2 (3)
Pyrexia (General disorders) | 5 (5) | 7 (7) | 8 (8) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Intermittent Rash Antecubital Fossae
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (13) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tooth Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pain due to broken tooth lower left jaw
Upper Respiratory Infection (Infections and infestations) | 1 (2) | 4 (5) | 3 (3) | 1 (1)
Upper Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Post Nasal Drip
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginitis Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Candidiasis (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Apthous Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Apthous Ulcer Buccal Mucosa
Blood Pressure Diastolic Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campbell de Morgan Spots (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Cherry Angioma Center Chest
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Chest Soreness
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Contact Dermatitis On Left Upper Arm
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 2 (3) — Sweats
Injection Site Erythema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Injection Site Hematoma (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Injection Site Pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Melanoicytic Naevus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Nevus in Pubic Area
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Left Wrist Strain
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (5) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No